CLINICAL TRIAL: NCT04257955
Title: COMMUNI.CARE (COMMUNIcation and Patient Engagement at Diagnosis of PAncreatic CAncer): Study Protocol
Brief Title: COMMUNIcation and Patient Engagement at Diagnosis of PAncreatic CAncer
Acronym: COMMUNICARE
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Gabriele Capurso, MD, PhD, Chief of Clinical Research, Pancreato-Biliary Endoscopy and Endosonography Division, Pancreas Translational and Clinical Research Centre, San Raffaele Scientific Institute, Milan, Italy, IRCCS San Raffaele
Other Study IDs: 51/INT/2019
Record Dates: First submitted 2020-01-31; First posted 2020-02-06 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Pancreatic Cancer; Interaction; Diagnosis
Keywords: doctor- patient interaction; pancreatic cancer; diagnosis communication
MeSH Terms: conditions — Pancreatic Neoplasms; Disease | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pancreatic cancer: Outpatients seen at the Gastroenterology, Pancreatic Surgery and Oncology Clinics of the Pancreas Translational and Clinical Research Centre, IRCCS San Raffaele, Milan (Italy) will be considered includable if:
  1. Adult patients (≥18 years);
  2. Of Italian mother tongue;
  3. Have a histologic diagnosis of PDAC obtained during the 4 weeks before the visit
  4. The visit is the first visit after completion of diagnostic procedures and is set to communicate the diagnosis and treatment strategies
  5. Give full, written informed consent
  The following exclusion criteria will be applied:
  1. PDAC recurrence after previous diagnosis and treatment
  2. poor performance status (ECOG ≥ 3);
  Interventions: Behavioral: Interview and evaluation of Engagement

INTERVENTIONS:
Behavioral: Interview and evaluation of Engagement — (i) the completion of the scheduled outpatients visit (ii) filling of the PHE-Scale® questionnaire by the patient to investigate the level of engagement and (iii) the completion of a semi-structured interview to assess the rate of understanding of the information received from the doctor.

SUMMARY:
BACKGROUND: The diagnosis of pancreatic adenocarcinoma (PDAC) in many cases is completely unforeseen by the patient, who often faces a disease that is already at an advanced stage, with poor prognosis. The clinical visit during which the diagnosis is communicated together with the first information regarding the planned treatments is of paramount importance. It is hypothesized that the clarity of such information is able to influence patients's engagement and thus the compliance.

AIMS: The aim of this study is to collect quantitative data on the level of PDAC patient engagement and the rate of understanding of the information received from the doctor, and investigate the possible association between these two variables and with the patient's level of compliance.

METHODS: This is a single-center, observational, cross-sectional cohort study focused on patients diagnosed with PDAC, approved by the Ethics Committee of the San Raffaele Hospital. As no preliminary data are available on the association between PDAC patient's understanding rate and their level of engagement and of compliance no power calculation is possible. This is a pilot study, aimed at enrolling at least 45 PDAC patients during a 3 months frame.

CONCLUSION: COMMUNI.CARE will be the first study specifically investigating whether there is a relation between PDAC patients' rate of understanding, their engagement and compliance at time of diagnosis.

DETAILED DESCRIPTION:
The diagnosis of PDAC in most cases is completely unforeseen for the patient, who faces with the disease already at an advanced stage and without a progressive approach to it. The clinical interview in which the diagnosis and the first information regarding treatment options and prognosis are communicated assumes a strong relevance, since it is an unexpected diagnosis with a poor prognosis.

Doctor-patient communication is an integral part of the care itself and poses the basis for the construction of the therapeutic alliance, an essential condition for compliance of the patient with reference to the treatments proposed by the physician.

Many recent studies claim that a good level of patient engagement is an essential condition for building a solid therapeutic alliance; in this regard, objective measurement scales of the patient engagement level have been developed, and have been demonstrated to be useful for quantifying the patient's involvement within the care process Among them is the Patient Health Engagement Scale (PHE-S®)-Scale, a recently validated assessment scale of simple and non-invasive use, that requires only the administration of a questionnaire to the previously informed patient who gives his consent.

The hypothesis of this study is that the clarity of the communication between the treating physician and the patient, and the level of understanding by the patient of the information conveyed by the doctor, in particular at the time of diagnosis largely influences the construction of a solid therapeutic alliance between the treating physician and PDAC patients and consequently the patient's engagement and compliance in the care process.

Our hypothesis is that the clarity of the communication between the treating physician and the patient and the degree of comprehension by the patient, especially during the first phases of the cure, are associated with the level of engagement and consequently with the compliance of patients with PDAC.

If the present pilot study will support the initial hypothesis, further action to improve the clarity of the clinical communication will be promoted.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years);
* Of Italian mother tongue;
* Have a histologic diagnosis of PDAC obtained during the 4 weeks before the visit
* The visit is the first visit after completion of diagnostic procedures and is set to communicate the diagnosis and treatment strategies
* Give full, written informed consent

Exclusion Criteria:

* PDAC recurrence after previous diagnosis and treatment
* Poor performance status (ECOG ≥ 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient (<18 years old), Italian mother tongue, enrolled during the visit that takes place at the time of the communication of the pancreatic cancer diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-04-19 (Actual)

PRIMARY OUTCOMES:
Patient Engagement Level | 3 months
  Patient Health Engagement Scale (PHE-S®)-Scale is a validated quantitative tool to measure engagement.
Patient's Rate of Understanding | 3 months
  a semi-structured interview of about 30 minutes to ask the patient questions concerning the clarity of the communication he had received from the doctor and the type of language used, to record the rate of understanding of the information will be employed to define whether the language used by the treating physician and its clarity for the patient allowed understanding defined as the rate.
Patient's Compliance | 6 months
  Defined as rate of therapies received compared to what was proposed and planned by the treating physicians.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Capurso, Principal Investigator — IRCCS San Raffaele
Locations (1):
- Gabriele Capurso, Milan, Italy